CLINICAL TRIAL: NCT05175443
Title: Surgeons Can Avoid Lasting Pain Through Exercise Literacy
Acronym: SCAPEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Uhl (Other)
Responsible Party: Sponsor-Investigator, Timothy Uhl, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 72626
Record Dates: First submitted 2021-12-14; First posted 2022-01-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Neck Pain; Shoulder Pain
Keywords: Surgeon
MeSH Terms: conditions — Neck Pain; Shoulder Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Repeated Measure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Intervention (Experimental): 1. Wall Angels:Stretching tight anterior shoulder musculature Participants will assume this position and slide their arms up and down the wall for 2 minutes.
  2. Cervical Spine Mobility: will be accomplished by having the participant stabilize their shoulders and side bend their head in various positions to stretch each side of their next for 2 minutes with 10-15 second holds in each position.
  3. Posterior shoulder strengthening: will be performed with shoulder externally rotating and squeezing the scapular with 5 second holds for 2 minutes.
  4. Thoracic Spinal mobility: to improve thoracic extension participants will use a strap or tennis ball and perform thoracic extension with 10 second holds for 2 minutes.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will be trained, by a physical therapist, to perform a set of four daily exercises requiring 1 sets of 2 minutes for each exercise totaling 8 minutes of targeted exercise per day for 8 weeks of the intervention. These exercises will be progressed or modified every 2-4 weeks to assure the participant is receiving maximal benefit for their exercise intervention.

SUMMARY:
The physical demands of surgery are in many ways similar to those of high-performance athletes. No professional athlete would consider performing without careful attention to strengthening and physical preparedness, yet surgeons routinely place rigorous demands on their bodies without any training plan specific to their work demands. A series of exercises were developed to help stretch and strengthen the key core muscles to support surgeons during operating to prevent neck pain. This study hypothesizes that Neck pain discomfort will decrease following an 8-week intervention program compared to baseline reported scores.

DETAILED DESCRIPTION:
Participant will be asked to fill out a series 5 questionnaires at beginning of the study, end of the 8-week intervention and 1 month later to determine how the exercise program affected their general health, neck pain, and function.

1. Demographic information about their age, height, weight, sex, surgical experience, surgical frequency, level of pain, and exercise frequency and types. (21 items)
2. A questionnaire about neck pain (10 items)
3. A questionnaire about how pain interferes with their life (8 items)
4. A questionnaire about general health (10 items)
5. A questionnaire about how much the participant typically exercise. (4 items) All these questionnaires can be completed on a computer or tablet and the data will be stored on a secure site (RedCap). This should be completed in approximately 20 minutes at each assessment.

Next participants will be instructed how to perform a series of 4 exercises described in the intervention

Every week the participant will be sent a 3-item questionnaire to report their level of pain, surgical burden, and exercise compliance for the week. There are only 3 multiple choice questions which should take approximately 1 minute to complete per week.

ELIGIBILITY:
Inclusion Criteria:

* must be an actively operating surgeon either faculty, fellow, or resident.
* Must report at least 4 out of 10 with pain at worst over the previous week at intake that is attributed to operating.

Exclusion Criteria:

* Participants will be excluded if they have prior neck or upper back surgery within the last year.
* If the participant has any other medical condition that would prevent the participant from performing shoulder and neck strengthening and stretching exercises.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index | Baseline, at end of 8 weeks of intervention
  The Neck Disability Index is 10 items, with each item consisting of likert type scale ranging from 0-4 with a lower score indicating less disability. The 10 items are summed for a total of potential 50 points which is then normalized to 100% scale by multiplying by 2.

SECONDARY OUTCOMES:
Worse Neck Pain | Baseline, at end of 8 weeks of intervention
  Numeric pain rating scale of worse pain for the week in the neck. Scale ranges from 0=no pain to 10=worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Tim L Uhl, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhusuny A, Cook M, Khalil A, Xie Y, Johnston V. Neck/Shoulder Problems and Visual Disturbances Among Surgeons: A Scoping Review. J Surg Res. 2020 Mar;247:413-428. doi: 10.1016/j.jss.2019.09.064. Epub 2019 Oct 31. PMID 31679800
- [Background] Daher A, Carel RS, Tzipi K, Esther H, Dar G. The effectiveness of an aerobic exercise training on patients with neck pain during a short- and long-term follow-up: a prospective double-blind randomized controlled trial. Clin Rehabil. 2020 May;34(5):617-629. doi: 10.1177/0269215520912000. Epub 2020 Mar 17. PMID 32183555
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Cleland JA, Childs JD, Whitman JM. Psychometric properties of the Neck Disability Index and Numeric Pain Rating Scale in patients with mechanical neck pain. Arch Phys Med Rehabil. 2008 Jan;89(1):69-74. doi: 10.1016/j.apmr.2007.08.126. PMID 18164333
- [Background] Lee PH, Macfarlane DJ, Lam TH, Stewart SM. Validity of the International Physical Activity Questionnaire Short Form (IPAQ-SF): a systematic review. Int J Behav Nutr Phys Act. 2011 Oct 21;8:115. doi: 10.1186/1479-5868-8-115. PMID 22018588